CLINICAL TRIAL: NCT01448018
Title: Pilot Study on Efficacy and Tolerance of Intravitreous Injection of Ranibizumab (Lucentis®) in Early-onset Central Retinal Vein Occlusion in Comparison to Hemodilution Using Erythrocytapheresis
Brief Title: Hemodilution Versus Ranibizumab in Early-onset Central Retinal Vein Occlusion
Acronym: CHIC-3
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Centre Hospitalier Intercommunal Creteil (Other)
Responsible Party: Principal Investigator, Agnes Glacet-Bernard, Principal Investigator, Centre Hospitalier Intercommunal Creteil
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2009-011403-23
Record Dates: First submitted 2011-09-29; First posted 2011-10-06 (Estimated); Last update posted 2014-08-13 (Estimated); Status verified 2014-08

CONDITIONS: Central Retinal Vein Occlusion
MeSH Terms: conditions — Retinal Vein Occlusion | interventions — Ranibizumab; Hemodilution

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- ranibizumab (Active Comparator): patients in this arm receive 3 monthly injection of ranibizumab
  Interventions: Drug: ranibizumab
- Hemodilution (Active Comparator): hemodilution using erythrocytapheresis is performed as early as possible after inclusion, in order to lessen hematocrit level (target hematocrit of 35%)
  Interventions: Procedure: hemodilution
- ranibizumab and hemodilution (Active Comparator): patients receive both treatments
  Interventions: Drug: ranibizumab; Procedure: hemodilution

INTERVENTIONS:
Drug: ranibizumab — 3 monthly intravitreous injection as soon as possible after the inclusion
  Other Names: Lucentis
  Arms: ranibizumab; ranibizumab and hemodilution
Procedure: hemodilution — hemodilution using erythrocytapheresis - target hematocrit: 35% - as soon as possible after the inclusion
  Arms: Hemodilution; ranibizumab and hemodilution

SUMMARY:
The purpose of this study is to compare ranibizumab injection to hemodilution at the early phase of Central Retinal Vein Occlusion (CRVO) and to determine if the combination of both treatments may have a synergic effect.

DETAILED DESCRIPTION:
Patients with recent-onset CRVO (lasting for less than 1 month)are randomly assigned to one of 3 groups: hemodilution using erythrocytapheresis alone, 3 monthly injection of ranibizumab alone, or both.

Patients are followed monthly during the 6-month study.

ELIGIBILITY:
Inclusion Criteria:

* CRVO confirmed by fluorescein angiography
* duration from onset of 1 month or less
* visual acuity of 20/32 or less

Exclusion Criteria:

* neovascular complication
* extensive retinal ischemia requiring prompt panretinal photocoagulation
* hematocrit level lower than 38%
* previous laser or surgery in the study eye, etc

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2010-01; Primary Completion 2013-06 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Change in visual acuity | 6 months
  Change in best-corrected visual acuity (ETDRS chart) between baseline and 6 months

SECONDARY OUTCOMES:
Gain in visual acuity of 2 ETDRS-lines or more | 6 months
  Number of patients who gained 2 lines or more between baseline and the 6-month visit

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Intercommunal Hospital, Créteil
  - Pitie-Salpetriere Hospital, Paris

REFERENCES:
- [Background] Glacet-Bernard A, Atassi M, Fardeau C, Romanet JP, Tonini M, Conrath J, Denis P, Mauget-Faysse M, Coscas G, Soubrane G, Souied E. Hemodilution therapy using automated erythrocytapheresis in central retinal vein occlusion: results of a multicenter randomized controlled study. Graefes Arch Clin Exp Ophthalmol. 2011 Apr;249(4):505-12. doi: 10.1007/s00417-010-1532-5. Epub 2010 Oct 17. PMID 20953877